CLINICAL TRIAL: NCT05200429
Title: Canadian Observational Study Evaluating the Long-term IMPACT of CFTR (Can-IMPACT CF)
Brief Title: Canadian Observational Study Evaluating the Long-term IMPACT of Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) Modulators on People With CF
Acronym: Can-IMPACT CF
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Rayment, Principle Investigator, University of British Columbia
Other Study IDs: H21-01707
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Cystic Fibrosis
Keywords: Trikafta; Cystic Fibrosis; CFTR Modulator Therapy; Respiratory Disease
MeSH Terms: conditions — Cystic Fibrosis; Respiration Disorders | interventions — elexacaftor, ivacaftor, tezacaftor drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Urine, Stool and Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pre-Therapy Participants: All CF people with CF who do not have any known contraindications to CFTR modulator therapy and will be initiated on CFTR modulator therapy by their treating physician as part of clinical care are eligible and will be asked to participate in this study.
  Interventions: Drug: Trikafta

INTERVENTIONS:
Drug: Trikafta — Highly Effective CFTR Modulator Therapy
  Other Names: Elexacaftor/Tezacaftor/Ivacaftor

SUMMARY:
This observational study intends to investigate health trends and data in cystic fibrosis patients all across Canada that are receiving modulator treatment so researchers can determine if CFTR treatments are effective over a long period of time and if so, which treatments work best for each individual. The study will collect clinical data from routine standard of care, patient reported outcomes via survey data and samples for a biobank.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed a CFTR modulator therapy and planning to commence modulator therapy within 30 days OR planning to switch modulator therapies within 30 days
* Participates in the Canadian Cystic Fibrosis Registry (CCFR)
* Informed consent by participant, or parent/legal guardian or assent

Exclusion Criteria:

* Known contraindications to CFTR modulator therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All people with CF who do not have any known contraindications to CFTR modulator therapy and will be initiated on CFTR modulator therapy by their treating physician as part of clinical care are eligible and will be asked to participate in this study
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To examine the long-term pulmonary and nutritional effects of CFTR modulators. | 5 years
To assess the long-term impact of CFTR modulators on patient-reported outcome measures including quality of life, disease burden, and physical activity. | 5 years
To establish a bio-repository to enable further investigations of the effectiveness of CFTR modulator therapies on biological markers and predictors of response. | 5 years
To establish the benefits of CFTR modulators compared to propensity-score matched historic CF populations followed in the Canadian CF registry. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Rayment, MDCM, Principal Investigator — University of British Columbia; Bradley Quon, MD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - St Paul's Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No